CLINICAL TRIAL: NCT02048891
Title: Ovulation Trigger With hCG Compared to GnRH Agonist in Patients With Repeated IVF Failures
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Rambam Health Care Campus (Other)
Responsible Party: Principal Investigator, Shahar Kol MD, Director, IVF Unit, Rambam Health Care Campus
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RMB-0427-13
Record Dates: First submitted 2014-01-27; First posted 2014-01-29 (Estimated); Results first posted 2015-06-08 (Estimated); Last update posted 2015-06-08 (Estimated); Status verified 2015-05

CONDITIONS: Infertility
MeSH Terms: conditions — Infertility | interventions — Triptorelin Pamoate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- hCG trigger (Active Comparator): Ovulation trigger with Ovitrelle 250 microgram, luteal support with vaginal progesterone: gel Crinone 8% daily.
  Interventions: Drug: hCG trigger
- GnRH agonist trigger (Experimental): ovulation trigger with Decapeptyl 0.2 mg, luteal support with 2 injections of 1,500 U hCG.
  Interventions: Drug: GnRH agonist trigger

INTERVENTIONS:
Drug: GnRH agonist trigger
  Other Names: Oovulation trigger with Decapeptyl 0.2 mg, luteal support with 2 injections of 1,500 U hCG.
  Arms: GnRH agonist trigger
Drug: hCG trigger
  Other Names: Ovulation trigger with Ovitrelle 250 microgram.; Luteal support with daily progesterone gel = Crinone 8%
  Arms: hCG trigger

SUMMARY:
Ovulation trigger is needed in in vitro fertilization (IVF) to get mature eggs. Routinely, human chorionic gonadotropin (hCG) is used for that purpose given its similarity to the natural hormone that does this job in a natural cycle (luteinizing hormone, LH). In a natural cycle another hormone takes part in the process (follicle stimulating hormone, FSH). To induce a natural-like ovulation surge that includes LH and FSH , gonadotropin releasing hormone (GnRH) agonist can be given.

The purpose of this study is to find out which approach may work better in IVF patients who experienced 4 IVF failures.

ELIGIBILITY:
Inclusion Criteria:

* IVF patients with at least 4 consecutive failures.
* On trigger day, no more than 10 follicles of 12 mm and up

Exclusion Criteria:

* History of moderate or severe OHSS.

Ages: 35 Years to 44 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 3 (Actual)
Dates: Start 2014-10; Primary Completion 2015-01 (Actual); Study Completion 2015-04 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- IVF Unit, Rambam medical Center, Haifa, Israel, Israel

RESULTS

PARTICIPANT FLOW:
Groups:
- hCG Trigger: Ovulation trigger with Ovitrelle 250 microgram, luteal support with vaginal progesterone: gel Crinone 8% daily.
  hCG trigger
- GnRH Agonist Trigger: ovulation trigger with Decapeptyl 0.2 mg, luteal support with 2 injections of 1,500 U hCG.
  GnRH agonist trigger
Period: Overall Study
Arm/Group | hCG Trigger | GnRH Agonist Trigger
Started | 2 | 1
Completed | 2 | 1
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | hCG Trigger | GnRH Agonist Trigger | Total
Number analyzed (Participants) | 2 | 1 | 3
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.5 (2.1) | 42 (0) | 41.7 (1.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 1 | 3
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Israel | 2 | 1 | 3

OUTCOME MEASURES:

1. Primary Outcome: Fetal Heart Activity 1 Month After Oocyte Retrieval
Description: Fetal heart activity as seen by vaginal ultrsound imaging 1 month after oocyte retrieval
Time Frame: 1 month after oocyte retrieval
Measure: Number; unit: participants with fetal heart activity
Arm/Group | hCG Trigger | GnRH Agonist Trigger
Number analyzed (Participants) | 2 | 1
participants with fetal heart activity | 0 | 0

2. Secondary Outcome: Patients Comfort During the Luteal Phase
Time Frame: During 2 weeks from day of oocyte retrieval
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | hCG Trigger | GnRH Agonist Trigger
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/1
Other Adverse Events (participants affected / at risk) | 0/2 | 0/1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes